CLINICAL TRIAL: NCT01725724
Title: Effects of the Sangvia Blood Collection System on Postoperative Infections in Orthopedic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009/763
Record Dates: First submitted 2012-04-17; First posted 2012-11-14 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2013-08

CONDITIONS: Coxarthrosis
Keywords: Autologous blood transfusion; Allogeneic blood transfusion; Infection rate
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Blood Transfusion, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allogeneic blood (Active Comparator): Allogeneic blood transfusion. Patients in this group will receive allogeneic red cell transfusions.
  Interventions: Procedure: Allogeneic blood transfusion
- Autologous blood (Experimental): Autologous blood transfusion. Patients in this arm will receive per- and postoperatively collected autologous blood collected with the Sangvia Blood Collection System. If teh amount of autologous blood is too small for the clinical need, additional allogeneic blood will be transfused.
  Interventions: Procedure: Autologous blood transfusion

INTERVENTIONS:
Procedure: Autologous blood transfusion — Per- and postoperative transfusion of autologous salvaged blood collected with the Sangvia Blood Collection System.
  Arms: Autologous blood
Procedure: Allogeneic blood transfusion — Transfusion of allogeneic blood according to the transfusion guidelines at each of the participating hospitals.
  Arms: Allogeneic blood

SUMMARY:
The purpose of this study is to compare the infection rate in patients receiving/not receiving their own blood, collected during surgery, during and after orthopedic surgery.

The hypothesis is that transfusion of autologous salvaged blood may reduce postoperative infection.

DETAILED DESCRIPTION:
Postoperative infections (both systemic and wound infections) are complications that should be avoided both due to the discomfort and the risk to the patients and for the corresponding increment of hospital costs.

There are some studies indicating that transfusion of autologous salvaged blood may reduce postoperative infections. This may be due to immunostimulating cytokines released in these products. However, as these cytokines also may cause adverse events as febrile transfusion reactions and activation of the complement and the coagulation cascades, the overall impact may be different.

There are two publications from an Austrian group indicating that allogeneic blood transfusion in orthopedic patients cause increased postoperative infection rate irrespectively of the leukocyte content of the red cell concentrates.

The Austrian studies were not randomized. Therefore, it would be useful to perform a randomized, prospective study where the patients receive transfusion of salvaged blood versus allogeneic red cell concentrate as their primary replacement product, respectively.

The purpose of the pilot study is to evaluate if transfusion of autologous salvaged blood reduces the infection rate in orthopedic patients compared with patients receiving allogeneic blood transfusion. The study is limited to one source of autologous blood; blood collected by the Sangvia Blood Collection System, and the study is partially sponsored by the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a risk of needing red cell transfusion after surgery estimated to be above 75%, judged by preoperative hemoglobin concentration and known risk of preoperative bleeding
* Patients over 16 years of age
* Patients who have consented to participate

Exclusion Criteria:

* Patients with a known hemolytic anemia (congenital or acquired)
* Patients for whom informed consent has not been obtained

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Body temperature | Participants will be followed for the duration of hospital stay, an expected average of 8 days.
  The body temperature is measured as a part of infection monitoring.
C-reactive protein (CRP) | Participants will be followed for the duration of hospital stay, an expected average of 8 days.
  CRP i measured as a part of infection monitoring. Because elevated CRP is expected after surgery it is necessary to measure other parameters to in order to monitor infection.
White blood cells (WBC) | Participants will be followed for the duration of hospital stay, an expected average of 8 days.
  WBC is measured and is a part of the infection monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Tor A Hervig, MD, PhD, Principal Investigator — Haukealnd University Hospital
Locations (4):
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Kysthospitalet i Hagevik, Hagavik
  - Soerlandet hospital, Kristiansand
  - Stord Hospital, Stord